CLINICAL TRIAL: NCT03771105
Title: The Impact of Phosphate Metabolism on Healthy Aging
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000023461; 1UL1TR001863-01 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hypophosphatemia; Rickets; Hypercalciuria; XLH; HHRH
MeSH Terms: conditions — Hypophosphatemia; Rickets; Hypercalciuria | interventions — Phosphates

STUDY DESIGN:
Masking Description: crossover parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Patients with hereditary hypophosphatemic rickets with HHRH (Experimental): Hereditary hypophosphatemic rickets with hypercalciuria (HHRH)
  Interventions: Drug: phosphate
- Patients with X-linked Hypophosphatemia (Active Comparator): Patients with X-linked hypophosphatemia
  Interventions: Drug: phosphate
- 15 Patients with X-linked Hypophosphatemia (Active Comparator): 15 Patients with X-linked Hypophosphatemia that will receive phosphate treatment for 30 days.
  Interventions: Drug: phosphate
- 15 Patients Hereditary hypophosphatemic rickets with HHRH (Active Comparator): 15 patients withHereditary hypophosphatemic rickets with hypercalciuria (HHRH) that will receive phosphate treatment for 30 days.
  Interventions: Drug: phosphate

INTERVENTIONS:
Drug: phosphate — The target daily phosphate (Pi) intake is 3,500 mg/day (dietary intake plus our supplementation) for this study. Subjects will take a supplement of Pi (as KPhos Neutral 250 mg/tablet) to reach this target. Subjects will receive treatment for 30 days.

SUMMARY:
Determine the association between duration and dose of chronic conventional therapy with Pi and renal (nephrocalcinosis/nephrolithiasis), vascular (endothelial function), and cardiovascular function (echo- cardiography) in patients with hereditary hypophosphatemic rickets with hypercalciuria (HHRH) and patients with X-linked hypophosphatemia (XLH).

DETAILED DESCRIPTION:
The central hypothesis of this proposal is that patients with X-linked hypophosphatemia (XLH), when matched for duration and dose of phosphate (Pi) therapy to patients with hereditary hypophosphatemic rickets with hypercalciuria (HHRH), will evidence greater cardiovascular and vascular debility than patients with HHRH. The overall objectives of this project are to utilize our existing longitudinal databases for individuals with XLH and HHRH through an interdisciplinary collaboration between pediatric and adult endocrinology to: i) quantify the impact of exposure to Pi therapy across the lifespan on cardiovascular and renal complications, which are key aging endpoints, ii) determine the acute response to Pi loading in XLH and HHRH by studying the changes in surrogate markers of cardiovascular and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Children above the age of 13 years
* Younger and older adults with XLH and HHRH with confirmed NPT2c mutations affecting both copies of the NPT2c gene (HHRH) or one copy of the PHEX gene (XLH)
* Be willing to provide access to prior medical records to determine eligibility including imaging, biochemical, medical, and surgical history data
* Be willing and able to complete all aspects of the study
* Be willing to adhere to the study visit schedule and comply with the assessments (in the opinion of the investigator).

Exclusion Criteria:

* Subjects will be excluded, if they are children younger than age 13 years
* Subjects that have other diseases likely to impact bone and mineral metabolism (e.g. renal, hepatic, gastrointestinal disorders, and malignancy),
* Subjects that are currently pregnant,
* Subjects that received medical therapy or developed any condition, which in the opinion of the investigator, could present a concern for either subject safety or difficulty with data interpretation.
* Subjects will be excluded from Aim 2, if they are unable to tolerate supplemental phosphate.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parathyroid Hormone (PTH) levels | 30 days
  PTH levels are expected to increase over baseline after phosphate supplement (Pi).
Fibroblast Growth Factor 23 (FGF23) levels | 30 days
  FGF23 levels are expected to increase over baseline after phosphate supplement (Pi).

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Bergwitz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03771105/ICF_000.pdf